CLINICAL TRIAL: NCT04057742
Title: AlloSure and AlloMap for the Monitoring of Antibody Mediated Processes After Kidney Transplantation
Brief Title: AlloSure for the Monitoring of Antibody Mediated Processes After Kidney Transplantation
Acronym: All-MAP
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); CareDx (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-0750; 1K23DK122136-01 (NIH); A534280 (Other: UW Madison); SMPH/MEDICINE/MEDICINE*N (Other: UW Madison); Protocol Version 3/13/2023 (Other: UW Madison)
Record Dates: First submitted 2019-08-13; First posted 2019-08-15 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Kidney Transplant Failure and Rejection
Keywords: Chronic Active Antibody Mediated Rejection; cAMR
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Participants have the option of banking blood and urine for the purpose of measuring inflammatory cytokines.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: 30 participants with a positive virtual crossmatch (VXM) at the time of transplant will be monitored for 12 months and undergo protocol biopsies on months 3 and 12 to detect subclinical rejection. Participants may also undergo clinically indicated biopsies for suspicion of rejection. AlloSure, AlloMap, immune cell phenotypes, and inflammatory cytokines will be measured at baseline (within 48 hours of transplant), 3 weeks, 6 weeks, 3 months (Standard of Care (SOC) biopsy), 6 months, 12 months (SOC biopsy), and additionally at the time of any indication biopsy (5-7 time points/participant). Participants in this group will be monitored for 12 months. Participants will be offered the option of donating either 22.5 mL of blood (Allosure+AlloMap+cytokines) or 52.5 mL of blood (Allosure+AlloMap+cytokines+immune cell phenotyping) at each visit. Participants may change their donation volume from 22.5 mL to 52.5 mL at any point during the study.
  Interventions: Diagnostic Test: AlloSure ddcfDNA assay; Diagnostic Test: AlloMap assay; Diagnostic Test: Inflammatory Cytokines; Diagnostic Test: Immune Cell Phenotypes
- Group B: 24 participants with De novo donor specific antibodies (dnDSA) will undergo a SOC biopsy within approximately three months to determine the incidence of Active Antibody Mediated Rejection (AMR). Immune cell phenotyping, AlloSure, and AlloMap will be measured at the time of the SOC biopsy (1 timepoint/patient). This is a single-time point study, unless participants are diagnosed with AMR and require treatment. In this case, they would be enrolled in group C (see below).
  Interventions: Diagnostic Test: AlloSure ddcfDNA assay; Diagnostic Test: AlloMap assay; Diagnostic Test: Immune Cell Phenotypes
- Group C: 15 additional participants with the diagnosis of Chronic Active Antibody Mediated Rejection (cAMR) will undergo standard of care therapy and be monitored for treatment response with a follow-up biopsy at three months. Immune cell phenotyping, AlloSure, and AlloMap will be used at baseline (prior to index biopsy) and 3 month (follow-up surveillance biopsy) (2 timepoints/participant). Participants in this group will be monitored per SOC for three months (time between the two biopsies).
  Interventions: Diagnostic Test: AlloSure ddcfDNA assay; Diagnostic Test: AlloMap assay; Diagnostic Test: Immune Cell Phenotypes

INTERVENTIONS:
Diagnostic Test: AlloSure ddcfDNA assay — 2.5 mL collection for Donor Derived Cell Free DNA at transplant, 3 weeks, 6 weeks, 6 months, 12 months post-transplant for Group A, at transplant for Group B, and transplant and 3 months for Group C
Diagnostic Test: AlloMap assay — 10 mL collection PAXgene blood sample at transplant, 3 weeks, 6 weeks, 6 months, 12 months post-transplant for Group A, at transplant for Group B, and transplant and 3 months for Group C
Diagnostic Test: Inflammatory Cytokines — 10 mL collection at transplant, 3 weeks, 6 weeks, 6 months, 12 months post-transplant for Group A
  Groups: Group A
Diagnostic Test: Immune Cell Phenotypes — Collection of up to 1 cup of urine for per participant each study visit

SUMMARY:
This is a prospective cohort observational study to assess the role of AlloSure Donor Derived Cell Free DNA (ddcfDNA) assay in the monitoring of three high-risk groups of kidney transplant patients for antibody mediated processes.

* Group A. Thirty participants with a positive Virtual Cross-Match (VXM) at the time of transplant will be monitored for 12 months
* Group B. Similarly, 24 participants with dnDSA will undergo a SOC biopsy within approximately three months to determine the incidence of Active Antibody Mediated Rejection (AMR)
* Group C. 15 additional participants with the diagnosis of Chronic Active Antibody Mediated Rejection (cAMR) will undergo standard of care therapy and be monitored for treatment response with a follow-up biopsy at three months

DETAILED DESCRIPTION:
This is a prospective cohort observational study to assess the role of AlloSure Donor Derived Cell Free DNA (ddcfDNA) assay in the monitoring of three high-risk groups of patients for antibody mediated processes.

The AlloSure assay will be combined with the AlloMAP assay (PAXgene blood sample); which is the first in history FDA-cleared genomic solid organ transplantation rejection blood test (AlloMap). Immune cell phenotypes and inflammatory cytokines will be examined. The combination of the three assays will provide a comprehensive molecular diagnostic and prognostic approach to antibody-mediated processes after renal transplantation. Additionally, formalin fixed paraffin embedded (FFPE) samples from kidney biopsies for subjects in all groups will be used to validate the nCounter platform. 3 slides from each biopsy will be sent to CareDx to be examined on the nCounter system. Other routine clinical data will be examined and assessed for correlation with the nCounter results. This will include AlloSure, Molecular Microscope, eGFR, creatinine, DSA as well as other key data fields taken from the Electronic Medical Record (EMR).

AlloMap Kidney is a lab-developed test and will be provided by CareDx, Inc. located at Brisbane, CA, and is designed, manufactured and used within a single CareDx laboratory. AlloMap Kidney is currently provided as "For Research use only" test and results are not intended for clinical diagnosis or patient management for "KidneyCare", which is the AlloSure-Kidney and AlloMap-Kidney tests combined.

* Group A. Thirty participants with a positive VXM at the time of transplant will be monitored for 12 months and undergo protocol biopsies on months 3 and 12 to detect subclinical rejection. Participants may also undergo clinically indicated biopsies for suspicion of rejection. AlloSure, AlloMap, immune cell phenotypes, and inflammatory cytokines will be measured at baseline (within 48 hours of transplant), 3 weeks, 6 weeks, 3M (SOC biopsy), 6M, 12M (SOC biopsy) and additionally at the time of any indication biopsy (5-7 time points/patient). Subjects in this group will be monitored for 12 months.
* Group B. Similarly, 24 participants with dnDSA will undergo a SOC biopsy within approximately three months to determine the incidence of AMR. Immune cell phenotyping, AlloSure and AlloMap will be measured at the time of the SOC biopsy (1 timepoint/patient). This is a single-time point study, unless participants are diagnosed with AMR and require treatment. In this case, they would be enrolled in group C (see below).
* Group C. 15 additional participants with the diagnosis of cAMR will undergo standard of care therapy and be monitored for treatment response with a follow-up biopsy at three months. Immune cell phenotyping, AlloSure and AlloMap will be used at baseline (prior to index biopsy) and 3M (follow-up surveillance biopsy) (2 timepoints/patient). Participants in this group will be monitored per SOC for three months (time between the two biopsies).

For all three groups, history and physical, blood draws and urine sample collections are performed per SOC. The only addition is blood sample collection and additional urine collection at the indicated SOC timepoints for AlloSure, AlloMap, immune cell flow cytometry, RNA-signatures, and inflammatory cytokines. In addition, leftover pathology slides that are stored in the pathology department will be sent out to CareDx for the purposes of performing the NanoString analysis. The slides will be returned to the pathology department after the NanoString analysis is complete.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipients (de novo or retransplant)
* Positive Virtual Crossmatch at transplant (Group A)
* Undergoing SOC biopsy for dnDSA (Group B)
* Proven cAMR (Group C)

Exclusion Criteria:

* Multi-Visceral transplant
* Contraindication to renal biopsy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney Transplant Recipients
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2024-04-07 (Actual); Study Completion 2024-04-07 (Actual)

PRIMARY OUTCOMES:
Incidence of Biopsy Confirmed AMR | up to 12 months post-transplant
  To determine whether AlloSure, immune cell phenotypes, and inflammatory cytokines predict the incidence of AMR, the outcome measure will be incidence of biopsy confirmed AMR. For participants with a positive virtual crossmatch (group A), protocol biopsies are performed at 3 and 12 months posttransplant. For participants with De novo donor specific antibodies (dnDSA) (group B), protocol biopsies are performed within 3 months.

SECONDARY OUTCOMES:
Banff Pathology | up to 3 months following initial diagnosis of cAMR
  To determine whether AlloSure and immune cell phenotyping predict the course of disease and/or response to treatment in participants with cAMR (Group C) the Banff pathology will be assessed.
Renal Allograft Function: Concentration of Serum Creatinine (sCr) | up to 3 months following initial diagnosis of cAMR
  To determine whether AlloSure predicts the course of disease and/or response to treatment in participants with cAMR, renal allograft function will be assessed by measuring sCR at baseline (index biopsy) and up to 3 months following SOC biopsy-proven cAMR.
Renal Allograft Function: Estimated Glomerular Filtration Rate (eGFR) | up to 3 months following initial diagnosis of cAMR
  To determine whether AlloSure predicts the course of disease and/or response to treatment in participants with cAMR, renal allograft function will be assessed by measuring eGFR at baseline (index biopsy) and up to 3 months following SOC biopsy-proven cAMR.
Renal Allograft Function: Urinary Protein to Creatinine Ratio (UPC) | up to 3 months following initial diagnosis of cAMR
  To determine whether AlloSure predicts the course of disease and/or response to treatment in participants with cAMR, renal allograft function will be assessed by measuring UPC at baseline (index biopsy) and up to 3 months following SOC biopsy-proven cAMR.
Percent of Biopsy Samples Measured on Nanostring nCounter That Validate Clinical Outcomes | experiment performed within 7 days of receiving sample
  Validation of Nanostring nCounter platform using FFPE kidney biopsy tissue to assess tissue GEP in the context of Allograft Rejection in Groups A, B, and C.
  GEP will be measured on the FFPE tissue to assess the patterns associated with allograft rejection. Samples will be retrospectively analysed from historic kidney biopsies performed, where the clinical diagnosis and outcome is known. Results will be compared to the gold standard of histopathology analysis.
Number of Genes Upregulated in Allograft Rejection | experiment performed within 7 days of receiving sample
  GEP analysis of FFPE tissue will be analysed to identify what pattern of genes are involved with different types of rejection and see whether the platform matches what has already been published in the literature.
Number of Genes Upregulated for BK Virus as determined by Nanostring nCounter | experiment performed within 7 days of receiving sample
  Genes within the Nanostring panel are associated with BK infection, will be examined with FFPE tissue taken from participants who had clinical BK infection.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Panzer, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin - Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Banff Foundation for Allograft Pathology — https://banfffoundation.org/

DOCUMENTS (1):
  • Informed Consent Form (2022-06-07): https://cdn.clinicaltrials.gov/large-docs/42/NCT04057742/ICF_000.pdf